CLINICAL TRIAL: NCT01234142
Title: A Phase 1, Investigator And Subject Blind (Sponsor Open), Randomized, Placebo Controlled, Parallel Cohort, Escalating Multiple Dose Study To Evaluate The Safety, Tolerability And Pharmacokinetics Of A Varenicline Transdermal Delivery System In Adult Smokers
Brief Title: A Study Evaluating the Absorption Of Varenicline Through The Skin Following Once Daily Application Of A Patch For 14 Days
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: A3051142
Record Dates: First submitted 2009-08-14; First posted 2010-11-04 (Estimated); Last update posted 2011-10-14 (Estimated); Status verified 2011-10

CONDITIONS: Smoking Cessation
Keywords: varenicline transdermal percutaneous transcutaneous transdermal delivery system patch
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 (Experimental)
  Interventions: Drug: varenicline free base patch
- Cohort 2 (Experimental)
  Interventions: Drug: varenicline free base patch; Drug: placebo patch
- Cohort 3 (Experimental)
  Interventions: Drug: varenicline free base patch; Drug: placebo patch
- Cohort 4 (Experimental)
  Interventions: Drug: varenicline free base patch; Drug: placebo patch

INTERVENTIONS:
Drug: varenicline free base patch — varenicline transdermal delivery system (12.0 mg payload [drug amount loaded in each patch]) will be applied to the skin once daily for 14 days
  Arms: Cohort 1
Drug: varenicline free base patch — varenicline transdermal delivery system (18.0 mg payload [drug amount loaded in each patch]) will be applied to the skin once daily for 14 days
  Arms: Cohort 2
Drug: placebo patch — Matched placebo transdermal delivery system will be applied to the skin once daily for 14 days
  Arms: Cohort 2
Drug: varenicline free base patch — varenicline transdermal delivery system (24.0 mg payload [drug amount loaded in each patch]) will be applied to the skin once daily for 14 days
  Arms: Cohort 3
Drug: placebo patch — Matched placebo transdermal delivery system will be applied to the skin once daily for 14 days
  Arms: Cohort 3
Drug: varenicline free base patch — 2 varenicline transdermal delivery systems (combined to achieve a maximum drug payload of 36 mg) will be applied to the skin, side by side once daily, for 14 days
  Arms: Cohort 4
Drug: placebo patch — Matched placebo transdermal delivery systems will be applied to the skin, side by side, once daily for 14 days
  Arms: Cohort 4

SUMMARY:
This study will evaluate the steady-state pharmacokinetics, safety and tolerability of a varenicline patch applied once daily to the skin for 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* male or female
* adult cigarette smokers of any race

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Subjects with active suicidal ideation or suicidal behavior within 1 year prior to Screening as determined through the use of the C-SSRS (Columbia-Suicide Severity Rating Scale) or active ideation identified at Screening or Day 0.
* Any condition possibly affecting drug absorption through the skin (eg, psoriasis).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2010-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve (AUC24); observed maximum plasma concentration (Cmax) in a given dosing interval and time of maximum plasma concentration (Tmax) | Days 1, 7 and 14
Observed accumulation ratio (Rac) | Days 7 and 14
Observed minimum plasma concentration (Cmin) in a given dosing interval, and peak: trough fluctuation (PTF) | Days 7 and 14
Terminal half life (t1/2) | Day 14-Day 19

SECONDARY OUTCOMES:
Dermal rating scores (as measured by the Rating Scale for Assessment of Application Site Dermal-Erythema, Edema and Irritation) | Days 1-14 (24 hpd); Days 1, 7-8 (1 and 12 hpd); Day 14 (1,6,12,24,48,72,96 and 120 hpd)
VAS scores for nausea (using a Visual Analog Scale) | Days 1-19 (daily)
Daily adhesion score (as measured by the Rating Scale for Adhesion) | Days 1-14 (12 and 24 hpd);Days 1, 7 and 14 (1 and 6 hpd)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Fargo, North Dakota, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3051142&StudyName=A%20Study%20Evaluating%20the%20Absorption%20Of%20Varenicline%20Through%20The%20Skin%20Following%20Once%20Daily%20Application%20Of%20A%20Patch%20For%2014%20Days